CLINICAL TRIAL: NCT03805438
Title: Determining the ED90 for Intrathecal 3% Chloroprocaine for Elective Cervical Cerclage Surgery
Brief Title: ED90 of 3% Chloroprocaine for Cervical Cerclage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00100699
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Results first posted 2021-09-01 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Cerclage, Cervical
MeSH Terms: interventions — chloroprocaine

STUDY DESIGN:
Intervention Model Description: Initial Patient (A#X) 45mg (1.5mL) of Chloroprocaine 3% (Nesacaine - Fresenius Kabi), will be drawn up into a 3 ml syringe (a 1 ml 'TB syringe' will be used to aspirate the drug in aliquots to ensure accuracy). The following additive will be added: 10 mcg (0.2ml) of fentanyl (50 mcg/ml) 0.3 ml of sterile 0.9% sodium chloride Thus the total volume in the syringe will be 2 ml. Study drugs will be prepared by one anesthesiologist (un-blinded) and administered by another anesthesiologist (blinded).
  Subsequent Patient (A#X+1) The dose of Chloroprocaine 3% based on outcome from prior subject and calculations mentioned previously will be added to 10 mcg (0.2ml) of fentanyl (50 mcg/ml). Sterile 0.9% sodium chloride will be added until the total volume in the syringe is 2 ml.
Masking Description: The solutions and their administration procedures are identical to those used outside this research and are almost exclusively used for patients requiring spinal anesthesia for cervical cerclage. The only deviation involves diluting the chloroprocaine with saline so that study solutions are of equal volume to maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chloroprocaine dose (Experimental): Initial Patient (A#X) 45mg (1.5mL) of Chloroprocaine 3% (Nesacaine - Fresenius Kabi), will be drawn up into a 3 ml syringe (a 1 ml 'TB syringe' will be used to aspirate the drug in aliquots to ensure accuracy). The following additive will be added: 10 mcg (0.2ml) of fentanyl (50 mcg/ml) 0.3 ml of sterile 0.9% sodium chloride Thus the total volume in the syringe will be 2 ml. Study drugs will be prepared by one anesthesiologist (un-blinded) and administered by another anesthesiologist (blinded).
  Subsequent Patient (A#X+1) The dose of Chloroprocaine 3% based on outcome from prior subject and calculations mentioned previously will be added to 10 mcg (0.2ml) of fentanyl (50 mcg/ml). Sterile 0.9% sodium chloride will be added until the total volume in the syringe is 2 ml.
  Interventions: Drug: Chloroprocaine Hcl 3% Inj

INTERVENTIONS:
Drug: Chloroprocaine Hcl 3% Inj — Initial Patient (A#X) 45mg (1.5mL) of Chloroprocaine 3% (Nesacaine - Fresenius Kabi), will be drawn up into a 3 ml syringe (a 1 ml 'TB syringe' will be used to aspirate the drug in aliquots to ensure accuracy). The following additive will be added: 10 mcg (0.2ml) of fentanyl (50 mcg/ml) 0.3 ml of sterile 0.9% sodium chloride Thus the total volume in the syringe will be 2 ml. Study drugs will be prepared by one anesthesiologist (un-blinded) and administered by another anesthesiologist (blinded).
  Subsequent Patient (A#X+1) The dose of Chloroprocaine 3% based on outcome from prior subject and calculations mentioned previously will be added to 10 mcg (0.2ml) of fentanyl (50 mcg/ml). Sterile 0.9% sodium chloride will be added until the total volume in the syringe is 2 ml.

SUMMARY:
The aim of this study is to identify the dose of intrathecal (IT) chloroprocaine that provides effective anesthesia in 90% of patients undergoing elective cerclage placement (intraoperative analgesic supplementation not required).

DETAILED DESCRIPTION:
Cervical cerclage is a procedure performed on pregnant women with cervical incompetence to reduce the risk of second trimester spontaneous abortion and preterm labor. This outpatient procedure is performed commonly under both general and regional anesthesia. In an effort to ensure rapid discharge some institutions prefer the use of general anesthesia; however, this has the disadvantage of exposing the fetus to general anesthetic drugs, increased risk of aspiration and a higher requirement for opioid analgesia post operatively. The benefits of neuraxial anesthesia for cerclage placement includes rapid onset of a dense sensory block, reduced fetus exposure to medications, and maintenance of maternal airway reflexes. Successful analgesia for cerclage placement requires a sensory block from S4-T10 dermatomes. Inadequate sensory coverage with a spinal anesthetic typically necessitates the conversion to general anesthesia adding risk to the mother and fetus while increasing intraoperative times and resources. Currently there are no studies determining optimum dose of spinal chloroprocaine for cervical cerclage. The investigators propose a dose determining study to determine the ED90 of intrathecal lidocaine and chloroprocaine which will help decrease incidence of inadequate anesthesia for cervical cerclage.

This is a multicenter, double blinded, dose ranging, biased-coin design study. Usual practice for regional anesthesia for cerclage placement consists of a mixture of 3% chloroprocaine and fentanyl. The exact dosing of the local anesthetic mixture used is dependent on the anesthesiologist's preference. Chloroprocaine provides a rapid onset of surgical anesthesia with little need for intraoperative analgesic supplementation. If there are contraindications for spinal anesthesia or patient refusal than general anesthesia is offered as an alternative.

The aim of this study is to assess the anesthetic quality of various doses chloroprocaine and in elective cerclage placement. Chloroprocaine is licensed and commonly administered intrathecally for cerclage placement.

To mitigate against the occurrence of inadequate analgesia in this ED90 study, a combined spinal-epidural technique will be utilized in order to provide supplemental analgesia via epidural top up if needed.

The investigators propose testing the hypothesis in patients scheduled for elective cervical cerclage placement. Participants will receive standard of care for anesthesia but in the context of a clinical trial with the addition of randomization, blinding, and more comprehensive evaluation of the trial outcomes (see outcomes objectives below).

The proposed study will be conducted over a 2 year period from January 2019 to September 2020.

Spinal Study Solutions The solutions and their administration procedures are identical to those used outside this research and are almost exclusively used for patients requiring spinal anesthesia for cervical cerclage. The only deviation involves diluting the chloroprocaine with saline so that study solutions are of equal volume to maintain blinding.

Initial Patient (A#X) 45mg (1.5mL) of Chloroprocaine 3% (Nesacaine - Fresenius Kabi), will be drawn up into a 3 ml syringe (a 1 ml 'TB syringe' will be used to aspirate the drug in aliquots to ensure accuracy). The following additive will be added: 10 mcg (0.2ml) of fentanyl (50 mcg/ml) 0.3 ml of sterile 0.9% sodium chloride Thus the total volume in the syringe will be 2 ml. Study drugs will be prepared by one anesthesiologist (un-blinded) and administered by another anesthesiologist (blinded).

Subsequent Patient (A#X+1) The dose of Chloroprocaine 3% based on outcome from prior subject and calculations mentioned previously will be added to 10 mcg (0.2ml) of fentanyl (50 mcg/ml). Sterile 0.9% sodium chloride will be added until the total volume in the syringe is 2 ml.

Rescue If the subject has discomfort and requests analgesia, then 5 ml of 3% chloroprocaine via the epidural route will be given, alternatively the anesthesiologist can treat the discomfort at his discretion. Other alternatives include intravenous fentanyl, ketamine, inhalational nitrous oxide and conversion to general anesthesia.

Riks/Benefit Risks of the procedure include the following: discomfort during placement (10% or 1 in 10), drop in blood pressure (1% or 1 in 100), headache (1% or 1 in 100), allergic reactions (0.001% or 1 in 100,000), bleeding or infection (0.001% or 1 in 100,000), damage to nerves (0.001% or 1 in 100,000), failure of the anesthetic or inadequate anesthesia and need for general anesthesia (0.1% or 1 in 1,000). The benefit of participating in the study is that perceived pain may be better controlled, however this cannot be guaranteed.

This study will be conducted at two study sites, the University of Arkansas for Medical Sciences in Little Rock, Arkansas and Duke University in Durham, North Carolina.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Singleton pregnancy
* ASA class II or III
* Cervical cerclage 1st or 2nd trimester of pregnancy
* Simple prophylactic cervical cerclage

Exclusion Criteria:

* Patient refusal
* Abdominal and complex cervical cerclage (e.g. bulging bag)
* BMI ≥ 50 kg/m2
* ASA class IV or above
* Contraindication to neuraxial anesthesia
* Allergy to chloroprocaine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 47 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Habib, MBBS, Principal Investigator — Duke University Hospital
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Duke University Hospital, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared between institutions insofar as it is required for the sequential study design when evaluating the primary outcome. The dose of chloroprocaine used for each procedure as well as the outcome of the surgery will dictate the dosing for the next patient at either institution. PHI will not be shared however.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study protocol will be shared between institutions and will be identical. The SAP, CSR, and analytic code is also shared and identical. The ICF however will be different and each institution will use its own version of the consent form.
Access Criteria: Shared data will be stored in REDCap to be used between institutions. The data will be shared by the PIs and all members listed on the Duke IRB submission both at Duke and UAMS. All statistical analyses will be done at Duke.

REFERENCES:
- [Derived] Sharawi N, Tan HS, Taylor C, Fuller ME, Landreth RA, Diomede OI, Williams M, Martinello C, Mhyre JM, Habib AS. ED 90 of Intrathecal Chloroprocaine With Fentanyl for Prophylactic Cervical Cerclage: A Sequential Allocation Biased-Coin Design. Anesth Analg. 2022 Apr 1;134(4):834-842. doi: 10.1213/ANE.0000000000005927. PMID 35139044

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chloroprocaine Dose
Started | 47
Completed | 45
Not Completed | 2
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
Age, Continuous [Mean (Full Range); unit: years] | 32 [29 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 14
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: The Dose of Intrathecal (IT) Chloroprocaine That Provides Effective Anesthesia in 90% of Patients Undergoing Elective Cerclage Placement (Intraoperative Analgesic Supplementation Not Required).
Description: Identification of the dose of intrathecal 3% chloroprocaine that will provide adequate anesthesia for a cervical cerclage to occur.
Time Frame: 60 minutes
Population: Participants who completed the study.
Measure: Number (95% Confidence Interval); unit: mg
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
mg | 49.5 [45.0 to 50.1]

2. Secondary Outcome: Maximum Pain Numerical Pain Rating Scale (NPRS) During Surgery (as Reported by Patient, Scored From 0-10 in the PACU).
Description: The scale from 0-10 is used where a score of 0 represents no pain at all and a score of 10 represents the worst pain a participant could imagine. It is reported as a single score at a single point in time. No subscales are used.
Time Frame: 60 minutes
Population: Participants who completed the study.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
score on a scale | 0 [0 to 0]

3. Secondary Outcome: Number of Participants Who Reported Nausea (Self-reported by Patient, Yes or no).
Description: Number of participants reporting nausea.
Time Frame: 60 minutes
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
Participants | 8

4. Secondary Outcome: Number of Participants With Observed Vomiting. (Observed Yes or no).
Description: Number of participants with observed vomiting.
Time Frame: 60 minutes
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
Participants | 1

5. Secondary Outcome: Number of Participants Reporting Itching. (Self-reported by Patient, Yes or no).
Description: Number of participants reporting itching.
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
Participants | 2

6. Secondary Outcome: Number of Patients Who Were Given Vasopressor Phenylephrine (and Ephedrine) BP Drops Greater Than 15% Below Baseline or < 100mg Hg Systolic.
Time Frame: 60 minutes
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
Participants | 13

7. Secondary Outcome: The Average Dose of Phenylephrine Given to Those Patients Whose BP Dropped Greater Than 15% Below Baseline or < 100mg Hg Systolic.
Description: All patients were analyzed for possible requirement of this intervention, though all participants did not require the intervention.
Time Frame: 60 minutes
Population: Participants who completed the study.
Measure: Mean (Inter-Quartile Range); unit: mg
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
mg | 320 [100 to 460]

8. Secondary Outcome: Overall Patient Satisfaction at Time of PACU Discharge.
Description: The scale used is 0-10 where 0 would represent completely unsatisfied and 10 would be completely satisfied. A 10 would imply that if a participant had to have the procedure performed again, it would be repeated in the exact same fashion it was carried out the first time. This will be assessed at the time of PACU discharge and will be asked one time. No subscales are used.
Time Frame: 60 minutes
Population: Participants who completed the study.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
score on a scale | 10 [10 to 10]

9. Secondary Outcome: Time to Resolution of Motor Block at End of the Cerclage Placement (Measured in the PACU).
Description: The motor block is assessed using the Bromage scale (1-5). The block is objectively assessed using this scale based on which joints a patient is able to mobilize following epidural or subarachnoid block. A score of 1 represents a patient who is unable to mobilize any lower extremity joint. A score of 5 represents a patient able to mobilize all lower extremity joints.
Time Frame: 60 minutes
Population: Participants who completed the study.
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
minutes | 60 [45 to 90]

10. Secondary Outcome: Time to Hospital Discharge as Measured as the Time Difference Between Local Anesthetic Injection and Discharge Time as Recorded in the Medical Notes
Time Frame: approximately 180 minutes
Population: Participants who completed the study.
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
minutes | 150 [139 to 186]

11. Secondary Outcome: Time From Spinal Block to Ambulation
Time Frame: up to 180 minutes
Population: Participants who completed the study.
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
minutes | 60 [45 to 90]

12. Secondary Outcome: Time From Spinal Block to Micturition
Time Frame: approximately 180 minutes
Population: Participants who completed the study.
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
minutes | 150 [139 to 186]

13. Secondary Outcome: Time to Complete Sensory Regression
Time Frame: up to 180 minutes
Population: Participants who completed the study.
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
minutes | 90 [75 to 105]

14. Secondary Outcome: Time to Resolution of Motor Block (Bromage Score of 5)
Description: as for outcome 9
Time Frame: up to 180 minutes
Population: Participants who completed the study.
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
minutes | 60 [45 to 90]

15. Secondary Outcome: Time to Readiness for PACU Discharge (Pre-defined Nursing Criteria)
Description: Readiness for PACU discharge would include a patient who is able to ambulate unassisted (indicating resolution of motor block), has vital signs within normal limits, has pain levels acceptable to the patient, and has been able to urinate.
Time Frame: approximately 180 minutes
Population: Participants who completed the study.
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Chloroprocaine Dose
Number analyzed (Participants) | 45
minutes | 150 [139 to 186]

ADVERSE EVENTS:
Time Frame: Approximately 180 minutes
Groups:
- Chloroprocaine Dose: Initial Patient (A#X) 45mg (1.5mL) of Chloroprocaine 3% (Nesacaine - Fresenius Kabi), will be drawn up into a 3 ml syringe (a 1 ml 'TB syringe' will be used to aspirate the drug in aliquots to ensure accuracy). The following additive will be added: 10 mcg (0.2ml) of fentanyl (50 mcg/ml) 0.3 ml of sterile 0.9% sodium chloride Thus the total volume in the syringe will be 2 ml. Study drugs will be prepared by one anesthesiologist (un-blinded) and administered by another anesthesiologist (blinded).
  Subsequent Patient (A#X+1) The dose of Chloroprocaine 3% based on outcome from prior subject and calculations mentioned previously will be added to 10 mcg (0.2ml) of fentanyl (50 mcg/ml). Sterile 0.9% sodium chloride will be added until the total volume in the syringe is 2 ml.
  At the completion of this study, there were no adverse events experienced by any patients enrolled in the study. As such, the delineation of adverse events on a per dose level is unnecessary.
Arm/Group | Chloroprocaine Dose
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT03805438/Prot_SAP_000.pdf